CLINICAL TRIAL: NCT06716892
Title: Non-invasive Preoperative Donor-site Evaluation of Free Flaps in Head and Neck Tumor Patients Using Multispectral Optoacoustic Tomography (MSOT)
Brief Title: Non-invasive Preoperative Tissue Evaluation in Head and Neck Tumor Patients Using Multispectral Optoacoustic Tomography (MSOT)
Acronym: msotcmfflap
Status: Recruiting | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: 24-335-B
Record Dates: First submitted 2024-11-29; First posted 2024-12-04 (Actual); Last update posted 2024-12-04 (Actual); Status verified 2024-11

CONDITIONS: Head and Neck Cancer; Healthy
Keywords: MSOT; Head and neck cancer; healthy; flap surgery; graft; perfusion; oxygenation
MeSH Terms: conditions — Head and Neck Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — whole blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Healthy: Healthy adult volunteers. Exclusion criteria: Chronical abuse of alcohol and nicotine, pregnancy and breastfeeding, ink / tattoo in the areas of interest (upper back, distal forearm, upper and lower leg)
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)
- Head and neck cancer patients.: Patients with histopathological diagnosed head and neck cancer.
  Interventions: Device: Multispectral Optoacoustic Tomography (MSOT)

INTERVENTIONS:
Device: Multispectral Optoacoustic Tomography (MSOT) — Non-invasive transcutaneous MSOT imaging of muscle and subcutaneos regions.

SUMMARY:
Multispectral Optoacoustic Tomography (MSOT) is a promising imaging technology that utilizes pulsed laser light. One of the key capabilities of this technology is measuring oxygenation within human tissue. This proposed study aims to investigate possible limitations of human tissue used for reconstructive surgery due to flawed tissue perfusion.

Healthy volunteers as well as patients with a diagnosed head and neck cancer entity will be recruited. Both cohorts will then be scanned on different body areas (most common tissue sites used for reconstructive surgery on the back, arms and legs) to assess differences in muscle oxygenation between the healthy and tumor patient cohort using MSOT.

The hypothesis of the study is, that patients with diagnosed head and neck cancer entities are prone to compromised tissue perfusion due to a high prevalence of smoking within the head neck tumor patient cohort and therefore perfusion restirciting diseases e.g. peripheral arterial occlusive disease (PAOD).

ELIGIBILITY:
Inclusion Criteria:

* Cohort 1: Histopathological diagnosed head and neck tumor patients.
* Cohort 2: Healthy adults.

Exclusion Criteria:

* Pregnancy / breastfeeding
* ink / tattoo in the areas of interest (upper back, distal forearm, upper and lower leg)
* missing consent form
* Cohort 2: Chronical abuse of alcohol and nicotine.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Eligible subjects are Histopathological diagnosed head and neck tumor patients of the cmf department of the University clinic of erlangen (1) and healthy volunteers who will be recruited from advertised announcements (2).
  All subjects meeting all inclusion and none of the exclusion criteria will be enrolled and added to their corresponding cohort (1 or 2).
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2024-11-28 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Muscle oxygenation (in arbitrary units) | Immediately before and after intervention (exercise) within both cohorts. Within the cohort of head and neck tumor patients, possible postoperative second measurement of the transplanted tissue after performed reconstructive surgery.
  Oxygenated hemoglobin signal in the measured muscle regions in all different cohorts.
Quantitative hemoglobin-associated signal (in arbitrary units) | Immediately before and after intervention (exercise) within both cohorts. Within the cohort of head and neck tumor patients, possible postoperative second measurement of the transplanted tissue after performed reconstructive surgery.
  Hemoglobin signal in the measured muscle regions in all different cohorts.

SECONDARY OUTCOMES:
Postoperative compromise of microvascular free flaps (Microvascular revision, flap failure) | Postoperative observation of the free flap within the stationary visit until dismission (14 days)
  Correlation between preoperative accquired MSOT parameters (e.g. quantitative hemoglobin-associated signal, muscle oxygenation, oxygen saturation) in the head and neck cancer cohort and the clinical outcome of the reconstructive surgery (Microvascular revision, flap failure).
Oxygen saturation (in %) | Immediately before and after intervention (exercise) within both cohorts. Within the cohort of head and neck tumor patients, possible postoperative second measurement of the transplanted tissue after performed reconstructive surgery.
  Proportion of oxygenated hemoglobin signal compared with total hemoglobin signal in the measured muscle regions in all different cohorts
Questionnaire items (Age, sex, height, weight, BMI, skin type, pre-existing conditions, medication, substance abuse [alcohol, nicotine], moderate physical activity per week) | Once at the date of inclusion for the study.
  Questionnaire items for both the healthy and the head and neck tumor cohort.
Muscle oxygenation (in arbitrary units) | Immediately before and after intervention (exercise) within both cohorts. Within the cohort of head and neck tumor patients, possible postoperative second measurement of the transplanted tissue after performed reconstructive surgery.
  Oxygenated hemoglobin signal in the measured muscle regions in all different cohorts.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Erlangen, Erlangen, Bavaria, Germany

IPD SHARING:
Plan to Share IPD: No
Due to the big amounts of acquired image data a publishing is not feasable.